CLINICAL TRIAL: NCT00286897
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Parallel Group Study of the Efficacy, Safety and Tolerability of E2007 in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Brief Title: The Efficacy, Safety and Tolerability of E2007 in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-E044-301; 2005-004314-33 (EudraCT Number)
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: E2007

SUMMARY:
Patients will be randomised to receive either placebo or the study drug for a period of 30 weeks, in addition to their standard Parkinsonian medications. During the first 8 weeks, the patient's levodopa doses may be adjusted if necessary by the investigator. For the remainder of the 22 weeks, all medications should be kept stable. Patients will be required to attend the clinic twice during the screening period and then a further 8 times during the treatment period. They will be required to complete home diaries where they will record their motor function. In addition, their doctor will assess their Parkinson's disease during the clinic visits. There will also be blood draws for safety and pharmacokinetic and pharmacogenomics evaluation. Following the treatment and assessment period, they will return to the clinic one month later for follow up.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female patients with idiopathic PD fulfilling the (UK) Parkinson's disease Society Brain Bank diagnostic criteria, with a good response to levodopa.
2. Patients must have been diagnosed with idiopathic PD at >= 30 years of age.
3. Patients must have predictable motor fluctuations of the wearing OFF type with the presence of at least 2 hours of OFF time during the waking day (excluding the morning OFF time) as evidenced by diary cards completed at screening and confirmed by diary data collected at the baseline visit.
4. Before patients are randomised they must be able to show that they are able to accurately complete the diary cards. During the diary-training period at the initial screening visit there must be diary evidence of at least one transition of OFF to ON or from ON to OFF and patients must show 75% concordance with Investigator's completion of the diary card.
5. Patients must rate between II-IV on the Hoehn & Yahr scale when in an OFF state.
6. Patients must be taking optimised levodopa therapy (according to investigator's opinion) at least 3 times during the waking day (not including bedtime/night time dose) up to a maximum of 8 doses daily (includes bedtime/night time dose).
7. Patients who are treated with dopamine agonists, COMT inhibitors or MAOB inhibitors and other anti-PD drugs must be on optimised and stable doses for at least 4 weeks prior to initial screening visit and must remain stable throughout the study. Only levodopa dosage can be adjusted downwards in the first 8 weeks of the double-blind treatment phase.
8. In the Investigator's opinion patients must be able to distinguish their own motor states and the absence or presence of troublesome or non-troublesome dyskinesias.
9. In the Investigator's opinion patients are able to complete the study including the completion of the home diary cards and capable of giving full written informed consent.

EXCLUSION CRITERIA:

1. Pregnant or lactating women.
2. Women of child bearing potential unless infertile (including surgically sterile) or practicing effective contraception (e.g., abstinence, IUD or barrier method plus hormonal method). These patients must have a negative serum B-HCG test at the initial screening visit (Visit 1), and a negative urine pregnancy test at the Baseline visit (Visit 3). These patients must also be willing to remain on their current form of contraception for the duration of the study. Postmenopausal women may be recruited but must be amenorrhoeic for at least 1 year to be considered of non-child bearing potential as determined by the investigator.
3. Fertile men not willing to use reliable contraception and fertile men with partners not willing to use reliable contraception.
4. Patients with a past or present history of drug or alcohol abuse as per DSM IV criteria.
5. Patients with a past (within one year) or present history of psychotic symptoms requiring antipsychotic treatment. Patients may be taking anti-depressant medication, however the dose must be stable for 4 weeks prior to the baseline visit. Use of anti-psychotic medication including clozapine and quetiapine is prohibited even if the indication is for movement disorders.
6. Patients with a past (within one year) or present history of suicidal ideation or suicide attempts.
7. Patients with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, gastro-intestinal, haematological, endocrine or metabolic systems which might complicate assessment of the tolerability of the study medication.
8. Patients with significantly elevated liver enzymes (abnormal bilirubin or serum transaminase levels of more than 1.5 times the upper normal limit).
9. Patients with current or prior treatment (within 4 weeks prior to the baseline visit) with medication known to induce the enzyme cytochrome P450 3A4.
10. Current or prior treatment (within 4 weeks prior to the baseline visit) with tolcapone, methyldopa, budipine, reserpine, seroquel or intermittent use of either liquid forms of levodopa or subcutaneous apomorphine.
11. Patients with previous stereotactic surgery (eg pallidotomy) for Parkinson's disease or with planned stereotactic surgery during the study period.
12. Patients receiving or with planned (next 6 months) deep brain stimulation.
13. Patients who have received an investigational product within 4 weeks prior to the screening visit or patients that have participated in a previous study with E2007.
14. Patients with clinically significant cognitive impairment (MMSE <24 and /or fulfilling DSM IV criteria for dementia due to Parkinson's disease).
15. Patients with conditions affecting the peripheral or central sensory system unless related to Parkinson's disease (such as mild sensory or pain syndromes limited to OFF periods) that could interfere with the evaluation of any such symptoms caused by the study drug.
16. Patients with any condition that would make the patient, in the opinion of the Investigator, unsuitable for the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2006-02; Primary Completion 2007-06 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Patient diaries: Change from baseline to final efficacy visit in the mean total daily OFF time (hr).

SECONDARY OUTCOMES:
Change from baseline on average OFF time over total treatment period; UPDRS Part II: OFF state; UPDRS Part III: ON state; change from baseline to final efficacy visit in mean total daily ON time w/o dyskinesias or with no troublesome dyskinesias.

CONTACTS AND LOCATIONS:
Overall Officials: Alessia Nicotra, MD, PhD, DIC, Study Director — Eisai Limited
Locations (118):
- Austria (2):
  - University Clinic Innsbruck, Innsbruck
  - Department of Neurology, Vienna
- Belgium (7):
  - Cliniques Universitaires St-Luc, Brussels
  - C.H.U.de Charleroi, Charleroi
  - U.Z. Antwerpen, Edegem
  - U.Z. Gent, Ghent
  - C.H.R. de la Citadelle, Liège
  - Hopital St-Pierre, Ottignies
  - St-Andries Ziekenhuis, Tielt
- Czechia (8):
  - University Hospital, Olomouc
  - University Hospital, Ostrava
  - Pliklinika Modry Pavilon, Ostrava
  - Nemocnice Pardubice, Pardubice
  - FN Plzen, Pilsen
  - Nemocnice Pisek, Plsek
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - VFN Praha, Prague
- Estonia (3):
  - Parnu Hospital, Pärnu
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- France (9):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Service Neurologie, Bayonne
  - CHU Gabrief Montpied, Clermont-Ferrand
  - Contis, Patrick, Colomiers
  - Lille
  - Centre de Pharmacologie Clinique et Evaluation Therapeutique, Marseille
  - Nantes
  - Hopital de la Pitie Salpetriere, Paris
  - Centre d'Investigation Clinique, Hospital Purpan, Toulouse
- Germany (16):
  - Kliniken Beelitz GmbH, Beelitz-Heilstätten
  - Uni-klinikum Charite, Campus Virchow-klinikum, Berlin
  - Bochum
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Neurologische Universitatsklinik, Göttingen
  - Universitatkrankenhaus Hamburg Eppendorf, Hamburg
  - Hanau
  - Hanover
  - Paracelsus-Elena-Klinik, Kassel
  - Gertrudis-Klinik, Parkinson Klinik, Leun-Biskirchen
  - Universitatsklinik Lubeck Klinik fur Neurologie Ratzeburger Allee 160 D-23538 Lubeck, Lübeck
  - Klinik fuer Neurologie, Marburg
  - Technische Universitaet Muenchen, München
  - LMU Munchen, Neurologische Universitatsklinik, München
  - Tübingen
  - Wiesbaden
- Hungary (10):
  - Clinexpert SMO, Budapest, Budapest
  - St. Imre Hospital, Budapest
  - Semmelweis University, Budapest
  - Uzsoki Street Hospital, Budapest
  - Jahn Ferenc Hospital, Budapest
  - B-A-Z County Hospital, Budapest
  - Budapest
  - A Petz Hospital, Győr
  - Nyiro Gyula Hospital, Győr
  - Jahn Ferenc Del-Pesti Hospital, Miscolc
- Israel (6):
  - Cham Sheba Medical Center, Haifa
  - Rabin MC, Petah Tikva
  - Ichilov Sourasky MC, Petah Tikva
  - Rambam Healthcare Center, Ramat Gan
  - Carmel Medical Center, Tel Aviv
  - Assaf Harofe Medical Center, Zerafin
- Italy (10):
  - Ospedal Villa Margherita, Arcugnano
  - Universita degli Studi di Genova, Genova
  - Ospedale della Misericordia, Grosseto
  - Policlinico Umberto I, Grosseto
  - Ospedale Versillia, Lido di Camaiore
  - Universita degli Studi Federico II, Napoli
  - IRCSS Fondazione Casimiro Mondino, Pavia
  - Ospedale Civile di Pescara, Pescara
  - Ospedale San Giovanni Battista, Roma
  - Roma
- Lithuania (3):
  - Kaunas Medical University Hospital, Kaunas
  - Vilnius University Emergency Hospital, Vilnius
  - Vilnius University Hospital, Santariskiu Clinic, Vilnius
- Poland (11):
  - Nzoz Kendrion, Bialystok
  - PSK Klinika Neurologii, Bialystok
  - Klinika Neurologii Doroslych AM, Gdansk
  - Centralny Szpital Kliniczny, Katowice
  - WSS im. Kardynala S. Wyszynskiego, Lublin
  - Lublin
  - Indywidualna Specjalistyczna Praktyka Lekarska, Gabinet Neur, Mosina k/Poznania
  - Specjalistyczna Przychodnia Lekarska, Płock
  - Centralny Szpital Kliniczny MSwia, Warsaw
  - Warsaw
  - Centrum Leczenia Chorob, Warsaw
- Portugal (3):
  - Servico de Neurologia, Coimbra
  - Hospital Santa Maria, Lisbon
  - Hospital Santo Antonio, Porto
- Serbia (3):
  - Clinic of Neurology and Psychiatry, Belgrade, Serbia and Montenegro
  - Clinic of Neurology, Belgrade, Serbia and Montenegro
  - Institute of Neurology, Belgrade, Serbia and Montenegro
- South Africa (10):
  - 407 Medi Clinic, Bloemfontein
  - Rosepark Hospital, Bloemfontein
  - Groote Schuur Hospital, Cape Town
  - Christian Barnard Memorial Hospital, Cape Town
  - 406 Claremont Hospital, Cape Town
  - Morningside, Johannesburg
  - Panorama Medi-Clinic, Parow
  - Wilgers Medical Centre, Pretoria
  - Sunninghill Hospital, Sunninghill, Johannesburg
  - Umhlanga Hospital, Umhlanga
- Spain (8):
  - Hospital Clinic I Provincial, Barcelona
  - Hospital de sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital del Mar, Servei de Neurologia, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
- Sweden (2):
  - Praktiken Ankaret, Karlstad
  - St Gorans Sjukhus, Stockholm
- United Kingdom (7):
  - Bupa Flyde Coast Hospital, Blackpool
  - North Surrey Primary Care Trust, Chertsey
  - District General Hospital NHS Trust, Clwyd
  - North Manchester General Hospital, Crumpsall
  - Royal Free Hospital, London
  - University College Hospital, London
  - Royal Hallamshire Hospital, Sheffield